CLINICAL TRIAL: NCT07286812
Title: Digital Technology Combined With Blood Marker Screening and Diagnosis for Community Populations Based on Classification Theory: an Integrated Study
Status: Not yet recruiting | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Liu Huayan, Neurology department, First Hospital of China Medical University
Other Study IDs: 2025733
Record Dates: First submitted 2025-11-26; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma and serum samples are retained and saved at -80 centigrade.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cognitive impairment group: The subjects diagnosed with AD-related cognitive impairment through early screening of cognitive disorders and examination of AD blood markers
- Healthy population group: The subjects who were diagnosed as negative through early screening for cognitive impairment and examination of AD blood markers

SUMMARY:
Our research hypothesis is as follows: A step - by - step screening strategy based on screening technologies can resolve the issue of insufficient efficiency in the traditional scale - based screening model. Meanwhile, performing pathological diagnoses on patients with suspected cognitive impairment identified through screening is conducive to the further implementation of etiology - based treatment and intervention, thus bringing benefits to patients at the earliest possible stage.

By exploring the characteristic changes in gait, facial expressions, and language of patients with suspected cognitive impairment and analyzing their diagnostic efficiency for cognitive impairment patients, new ideas can be provided for the early diagnosis of the disease.

Through longitudinal observation of the changes in disease - related information during the progression and transformation of the disease, a predictive model for the early diagnosis of cognitive impairment and the prediction of disease progression can be constructed.

DETAILED DESCRIPTION:
Cognitive impairment refers to the impairment of cognitive functions caused by various factors, involving multiple cognitive domains such as orientation, memory, calculation ability, attention, language function, executive function, reasoning ability, and visuospatial function, and affecting patients' social functions and quality of life to varying degrees. Cognitive impairment is classified into mild cognitive impairment and dementia based on its severity. Alzheimer's disease is the most common type of dementia causing cognitive impairment, accounting for 60% to 80% of all dementia cases. The prevalence of cognitive impairment is increasing rapidly and showing a trend of younger onset, becoming a pressing public health issue in the process of global aging.

Dementia in the elderly, especially Alzheimer's disease, generally undergoes a 15 to 20-year latent development process. Studies have shown that through early screening to identify high-risk individuals and implement precise intervention, the rate of cognitive decline can be effectively reduced, and the disease progression can be delayed. Communities, as the main place for the elderly's daily life, are important platforms for implementing dementia screening and health intervention. Conducting early screening in the community population and adopting a forward-looking prevention strategy can effectively identify patients at the stage of mild cognitive impairment. Through comprehensive intervention measures such as improving lifestyle, controlling chronic diseases, and strengthening cognitive training, the occurrence and development of cognitive impairment can be effectively prevented or delayed. For identified dementia patients, establishing an effective multi-level cognitive impairment prevention and intervention system "hospital - community - family - patient" will help improve the quality of life of patients. Early screening and diagnosis of cognitive impairment is extremely important, and researching the early screening and diagnosis system of cognitive impairment is of great significance.

How to improve the ability of cognitive impairment screening tools, optimize the diagnostic process, has always been a key scientific issue in establishing a cognitive impairment early screening and diagnosis system. Studies have found that through a two-stage stratified screening scheme combining rapid pre-screening with AMT/PFQ and precise diagnosis with MMSE/MOCA, the screening time can be shortened by more than 50%, and the negative predictive value remains above 99%. This optimized path reduces the cost consumption in the resource-intensive stage by shrinking the scale of individuals requiring advanced cognitive assessment. Moreover, the latest research shows that many clinical symptoms of AD occur in the early stage of the disease, which can not only help indicate the occurrence of the disease but also help predict the progression of the disease. However, these symptoms are often complex and difficult to be comprehensively and accurately evaluated through clinical observation by doctors, such as gait abnormalities, facial expressions, and language disorders. Gait is a very complex task that requires coordinated interaction of a wide range of brain regions to complete, and mild cognitive impairment will lead to abnormal gait. Therefore, gait abnormalities not only reflect the severity of dementia but also can help indicate early mild cognitive impairment and predict the occurrence of cognitive impairment. Existing research on the assessment of gait abnormalities still relies on quantitative indicators such as walking speed, stride length, and stride width, but gait is a dynamic process, and these indicators cannot comprehensively and precisely reflect the overall situation of gait abnormalities of patients. The olfactory cortex is most easily damaged in the early stage of AD, and the damage of the amygdala will specifically lead to the disorder of emotion processing in patients, especially the disorder of facial expression recognition and expression. More research indicates that the disorder of emotion recognition and expression will seriously affect the quality of life of patients and is the main reason for conflicts and burdens between caregivers and patients. However, there is still less research on facial expression disorders, and there is no effective method for identifying and evaluating the abnormality of patients' facial microexpressions and their emotional perception disorders. Language disorder is the core feature of cognitive impairment, which not only can predict the occurrence of cognitive impairment but also can reflect the severity of cognitive damage. However, there is still no universal system in clinical practice for comprehensive detection of language disorders. Currently, it mainly relies on specialist doctors using various complex scales to assess patients' language disorders. This often leads to significant differences in symptom assessment and interpretation. In summary, gait, facial expressions, and language disorders can all play important roles in the early diagnosis and disease course assessment of AD and MCI.

Our research hypothesis is: The stepwise screening strategy based on screening techniques can solve the problem of insufficient efficiency in the traditional scale screening model. At the same time, conducting pathological diagnosis for suspected cognitive impairment patients can help further implement etiological-based treatment and intervention, bringing benefits to patients as early as possible; by exploring the change characteristics of gait, facial expressions, and language in suspected cognitive impairment patients, analyzing their diagnostic efficacy for cognitive impairment patients, providing new ideas for early diagnosis of the disease; through longitudinal observation of the changes in disease-related information as the disease progresses and transforms, constructing a prediction model for early diagnosis and disease progression of cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 50 and above;
2. Residents of this community for at least one year, with established medical records;
3. Deny a history of cognitive impairment diseases (mild cognitive impairment, dementia, Alzheimer's, etc.) and the use of anti-dementia drugs (cholinesterase inhibitors or memantine, etc.);
4. Agree to participate in the study;
5. The individual and their relatives can communicate normally in Chinese.

Exclusion Criteria:

1. Self-reported or confirmed through inquiry that there is a severe mental disorder, such as bipolar disorder or schizophrenia, etc.
2. Suffering from a disease that makes it impossible to complete the cognitive assessment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents aged 50 and above who were included in the communities from December 2025 to April 2026
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic efficiency of the cognitive impairment screening and diagnosis protocol | 1 year
  The diagnostic efficiency will be measured by the area under curve（AUC）of receiver operating characteristic（ROC）curve.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 12 months after publication
Access Criteria: the IPD and any additional supporting information will be shared with the researchers who follow our idea and theory, and concern on the AD and MCI diagnosis. Huayan Liu will review the requests.